CLINICAL TRIAL: NCT03705026
Title: Relationship Between Genetic Polymorphism and Postoperative Nausea and Vomiting Undergoing Breast Surgery With General Anesthesia in Chinese Han Population
Brief Title: Relationship Between Genetic Polymorphism and Postoperative Nausea and Vomiting in Chinese Han Population
Status: Completed | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UnionAnesthesia
Record Dates: First submitted 2018-10-06; First posted 2018-10-15 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2018-10

CONDITIONS: Breast Neoplasms; Anesthesia, General
Keywords: postoperative nausea and vomiting; general anesthesia; breast surgery; single nucleotide polymorphism
MeSH Terms: conditions — Breast Neoplasms; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with whole blood DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative nausea and vomiting ( PONV ) is one of the common complications after general anesthesia while genetic factors may play an important role in Postoperative nausea and vomiting. In this study, the investigators investigated the relationship between gene polymorphism ( such as single nucleotide polymorphism ) of the gene HTR3A ( 5-hydroxytryptamine receptor 3A ), HTR3B ( 5-hydroxytryptamine receptor 3B ), HTR3C ( 5-hydroxytryptamine receptor 3C ) and TACR1 ( tachykinin receptor 1 ) etc. with nausea and vomiting after general anesthesia. Simultaneously, the investigators explored the influencing factors of nausea and vomiting.

DETAILED DESCRIPTION:
Materials and methods:

Demographic data and risk factors responsible for PONV, including the history of PONV and motion sickness, were collected preoperatively by interviewing participants the day before anesthesia.

All study subjects received a standardized anesthesia regimen. General anesthesia was induced by midazolam 0.04 mg/kg, propofol 1.5 mg/kg, sufentanil 0.4 μg/kg, and cisatracurium 0.2 mg/kg (to facilitate tracheal intubation) given intravenously.Participants' lungs were ventilated with 50% oxygen in air.

During general anesthesia, concentration of sevoflurane maintained 1.0% to 3.0% at the discretion of anesthetist who was not involved in the study. General anesthesia also uses propofol 1 mg kg-1 h-1 and sufentanil 0.1 μg kg-1 h-1 by continuous intravenous infusion. An Entropy index monitor was used to maintain the appropriate anesthesia depth by 40-60. Participants received a repeated bolus of sufentanil 0.1 μg/kg or cisatracurium intravenously on demand.

After surgery the investigators recorded the data such as Anesthesia duration, doses of sufentanil and propofol and so on.

At the end of surgery and after returning to the ward, flurbiprofen axetil 50 mg injection i.v. was administered as an analgesic therapy, respectively. Cholinesterase inhibitor-based neuromuscular reversal drugs and vitamine B6 were not administered after surgery. Bucinnazine hydrochloride 100 mg intramuscular injection (i.m.) as a rescue medication was administered to any participant whose visual analogue scale/score (VAS) was > 3.

Ondansetron was given intravenously to the participants if necessary or requested . Unaware of the genotypes of the subjects, the investigators collected the participants' data including nausea, vomiting and pain.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing breast surgery with general anesthesia
* American Society of Anesthesiologists Physical Status Classifications 1-2
* No history of smoking
* body mass index (BMI) <35 kg/m2

Exclusion Criteria:

* Declined to participate
* Had used antiemetics, steroids, H2 antagonists, anticholinergics, antihistamines, butyrophenones, phenothiazines, metoclopramide or opioids within 24 hours
* Gastroesophageal reflux, gastrointestinal obstruction or ulcer, vestibular or hearing dysfunction
* Liver impairment, renal impairment, psychiatric disorder, chronic pain
* Pregnant and lactating patients
* Requiring postoperative patient-controlled analgesia
* Requiring prophylactic use of antiemetics
* Allergic to drugs related in the study
* Receiving chemotherapy within one week before surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Han population who were admitted to department of breast surgery, Fujian Medical University Union Hospital.
Sampling Method: Probability Sample
Enrollment: 568 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Whether the participants occur nausea or not | Period of 0 to 6 hours after surgery
  Nausea was defined as a feeling of wanting to throw up or about to throw up.
Whether the participants occur vomiting or not | Period of 0 to 6 hours after surgery
  Vomiting was defined as the discharge of the stomach contents, while retching as an involuntary attempt to vomit that did not produce stomach contents. Retching was considered as vomiting.
Whether the participants occur nausea or not | Period of 6 to 24 hours after surgery
  Nausea was defined as a feeling of wanting to throw up or about to throw up.
Whether the participants occur vomiting or not | Period of 6 to 24 hours after surgery
  Vomiting was defined as the discharge of the stomach contents, while retching as an involuntary attempt to vomit that did not produce stomach contents. Retching was considered as vomiting.

SECONDARY OUTCOMES:
Level of nausea | Within 24 hours after surgery
  The level of participants' nausea was rated on four-point scales: 0=no nausea; 1=mild nausea with activities; 2=mild nausea at rest; and 3=se-vere nausea at rest.
Number of vomiting | Within 24 hours after surgery
  The investigators defined an emetic episode as a single occurrence of vomiting/retching or as a series of immediately successive vomiting/retching. However, vomiting/retching had to be separated by at least 1 minute to be classified as a single emetic episode.

CONTACTS AND LOCATIONS:
Overall Officials: Liangcheng Zhang, Ph.D, Principal Investigator — Fujian Medical University Union Hospital

REFERENCES:
- [Derived] Yan T, Su J, Zhou L, Zhang L. Polymorphisms of 5-hydroxytryptamine receptor type 3B gene and clinical characteristics for vomiting after breast surgery in chinese han female population. J Clin Pharm Ther. 2021 Aug;46(4):936-941. doi: 10.1111/jcpt.13386. Epub 2021 Feb 19. PMID 33605481